CLINICAL TRIAL: NCT04090346
Title: Fecal Microbiota Transplant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 010.GID.2018.A
Record Dates: First submitted 2019-08-12; First posted 2019-09-16 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2021-11

CONDITIONS: Clostridium Difficile Infection
Keywords: CDiff; Fecal Microbiota Transplant; Infection Control; Antibiotic Stewardship
MeSH Terms: conditions — Clostridium Infections | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Clostridium difficile infection (Experimental): Clostridium difficile infection (CDI) is due to a toxin-producing bacteria that causes a more severe form of antibiotic associated diarrhea. The disease ranges from mild diarrhea to severe colon inflammation that can even be fatal.
  Interventions: Drug: Fecal Microbiota Transplant

INTERVENTIONS:
Drug: Fecal Microbiota Transplant — Fecal Microbiota Transplant (FMT) is a procedure to replace beneficial bacteria which has been killed or suppressed in the colon.
  Other Names: FMT

SUMMARY:
The study will provide data to show the effectiveness of Fecal Microbiota Transplant in patients with recurrent Clostridium difficile infection.

Fecal Microbiota Transplant (FMT) is a procedure in which healthy colon contents of a carefully screened donor is inserted into the colon of a compromised patient. FMT is a procedure to replace beneficial bacteria that has been killed or suppressed, most commonly by use of antibiotics. Currently it is utilized as an experimental treatment for Clostridium difficile infection (CDI). This procedure is predicted to reduce the cost both financially and physically for the CDI patient and facility.

DETAILED DESCRIPTION:
Methodist Health System wishes to offer transplant services to our CDI populations which meet all criteria for recurrent intractable disease. The objective is to reduce the cost both financially and physically to patients and the facility, of living with chronic or recurrent CDI disease. This study is to provide treatment and demonstrate documented outcomes and success rates in a manner that protects both the patients and the facility. Of note this treatment is currently being provided by many facilities in Texas, under the FDA Investigational New Drug (IND) enforcement discretion.

The study will provide data to show the effectiveness of Fecal Microbiota Transplant in patients with recurrent Clostridium difficile infection. This study will only examine FMT as it is the only available therapy beyond antibiotic treatment. When patients are considered for FMT they have already failed traditional therapeutic medications.

Patients will be required to meet a specified criteria set forth for chronic or severe CDI infection. Chronic infection is defined as the third or greater episode of C Difficile infection, proven by a positive stool assay with previous documented treatments. Patients must be first treated with first line drug therapies which include vancomycin, metronidazole or fidaxomicin without cure. They must have been treated with at least one course of drugs over a six to eight week period of a vancomycin taper or vancomycin treatment followed by rifaximin for two weeks. Severe CDI infection is defined as refractory moderate to severe CDI diarrhea, with failing vancomycin drug therapy.

Patients with contraindicated co-morbidities will be excluded. Comorbidities include severe bowel disease which would preclude colonoscopy, severe underlying immune suppression or decompensated liver cirrhosis.

Patients will be under the care of a physician who is an identified investigator (sub-investigator) of this study for preparation, procedure and follow up care. Patients will be counseled by this physician regarding the risks and side effects of the procedure and transplant. Staff will only reinforce details from written materials given to patients. Questions outside of the written materials will be directed to the investigators for follow up.

Risks include, but are not limited to the following.

* Transplant making no improvement in the course of their CDI.
* Common side effects including transient gas, bloating and rectal irritation
* Surgical risks which can include blood clots, excessive bleeding, allergic reactions and death. More common surgical risks are infection, drug reactions, bleeding, and perforation.
* Transmission of antibiotic-resistant bacteria: These are resistant to one or more antibiotics. These bacteria could be transmitted through FMT and cause a serious infection. The FMT that you will receive is provided by a company called OpenBiome, where donors who provide stool for the FMT treatments undergo screening for certain antibiotic-resistant bacteria and clinical risk factors that would make their exposure to antibiotic resistant bacteria more likely. Individuals who test positive for these bacteria or have these risk factors are excluded from donating.

Patients will sign three informed consents. The first consent is to acknowledge the basis of the treatment is part of a research study (exhibit 1). The second consent) specifies that FMT is experimental in nature, and reviews the potential risks and benefits of the transplant. The third is the Methodist Health System "Disclosure and Consent" that is used for colonoscopy procedures.

ELIGIBILITY:
Inclusion Criteria:

* Recurring CDI after three episodes of mild to moderate C Diff infections and failure to respond to appropriate antimicrobial treatment of six to eight weeks.
* Metronidazole
* Vancomycin
* At least two episodes of severe C diff infection that have required hospitalization and significant morbidity within one year
* Severe C Diff infection requiring hospitalization and non- responsive to maximal medication therapy

Exclusion Criteria:

* advanced Human Immunodeficiency Virus (HIV) or Acquired Immunodeficiency Syndrome (AIDS)
* cirrhosis of the liver
* recent bone marrow transplants
* medication suppressed immune systems (allowed per physician discretion if benefit outweighs risk)
* pregnancy
* Toxic megacolon or ileus present

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
treatment date | eight weeks following transplant.
  date of treatment
material volume | eight weeks following transplant.
  volume of material
severity and type of CDI | eight weeks following transplant.
  severity and type of CDI
serious adverse reactions | eight weeks following transplant.
  serious adverse reactions
repeat transplant, colectomy and antibiotics | eight weeks following transplant.
  patients who require additional treatment

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Memon, MD, Principal Investigator — Methodist Mansfield Medical Center
Locations (1):
- Methodist Mansfield Medical Center, Dallas, Texas, United States